CLINICAL TRIAL: NCT00259298
Title: The Use of Nuclear Scintigraphy to Evaluate the Anabolic Effects of Teriparatide on the Skeleton in Postmenopausal Women With Osteoporosis
Brief Title: Evaluation of the Effects of Teriparatide on Skeleton Images in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9917; B3D-US-GHCV (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Results first posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Teriparatide (Experimental): Participants receive teriparatide 20 microgram once daily by subcutaneous injection for 18 months followed by 6 months off therapy
  Interventions: Drug: teriparatide

INTERVENTIONS:
Drug: teriparatide — Subcutaneous, 20 microgram (mcg)/day, 18 months
  Other Names: LY333334; Forteo; Forsteo

SUMMARY:
The purpose of this study is to evaluate the effects of teriparatide on skeleton images in postmenopausal women with osteoporosis. Teriparatide is a bone formation agent that stimulates the production of new bone in the skeleton. This process of bone formation can be studied using a technique commonly referred to as a bone scan or nuclear scintigraphy. This trial will test whether bone scans will identify areas of the skeleton that are forming new bone during teriparatide therapy. It also will study what these areas look like after therapy is stopped.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory with osteoporosis
* Hip or spine bone mineral density (BMD) measurement more than 2.5 standard deviations below the average bone mass of young healthy women or more than 2.0 standard deviations in women who have a history of a vertebral or nonvertebral fragility fracture.

Exclusion Criteria:

* Diseases of bone other than osteoporosis
* Treatment with estrogens in the 3 months prior to enrollment or for more than 2 months in the past year
* Treatment with oral bisphosphonates in the 3 months prior to enrollment or for more than 2 months in the past year; treatment with intravenous bisphosphonates in the 12 months prior to enrollment
* Increased risk for the development of osteosarcoma

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, London, United Kingdom

REFERENCES:
- [Derived] Moore AE, Blake GM, Taylor KA, Rana AE, Wong M, Chen P, Fogelman I. Assessment of regional changes in skeletal metabolism following 3 and 18 months of teriparatide treatment. J Bone Miner Res. 2010 May;25(5):960-7. doi: 10.1359/jbmr.091108. PMID 19929434
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Teriparatide: Participants received teriparatide 20 microgram once daily by subcutaneous injection for 18 months, followed by 6 months off therapy
Period: Overall Study
Arm/Group | Teriparatide
Started | 12
Received at Least 1 Dose of Study Drug | 10
Completed | 9
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Teriparatide
Number analyzed (Participants) | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 67.17 (7.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 12
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12
Qualitative Visual Assessment of Diffuse Uptake of 99m Technetium methylene diphosphonate [Number; unit: participants] — Presented are data only for participants who received a bone scan at baseline. Initial bone scans for each participant were evaluated by a radiologist for an increase in diffuse uptake in the whole skeleton compared to expected values in a healthy population. Subjective visual assessment categorized results into no increase, possible increase, and definite increase.
  participants
    no increase | 10
    possible increase | 0
    definite increase | 0
    not assessed | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kg/m2 | 24.56 (5.16)
Height [Mean (Standard Deviation); unit: centimeter] | 161.25 (6.88)
Qualitative Visual Score of Focal uptake of 99m Technetium methylene diphosphonate (99m Tc-MDP) [Mean (Standard Deviation); unit: units on scale] — Changes in focal uptake (localized, defined areas of uptake) in the whole skeleton were visually scored. Changes were rated on a scale from 0-4: 0=no clinically significant focal areas of skeletal uptake; 1=focal areas affecting <1% of skeleton; 2=focal areas affecting >=5% of skeleton; 3=focal areas affecting >=20% of skeleton; 4=focal areas affecting >=50% of skeleton.
  units on scale | 0.7 (0.48)
Skeletal plasma clearance of 99m Technetium methylene diphosphonate (99m Tc-MDP) [Median (Inter-Quartile Range); unit: milliliter/minute] — Skeletal plasma clearance is defined as the volume of plasma cleared of tracer (99m Tc-MDP) by the skeleton per unit time (milliliter/minute). Kbone is the rate constant representing plasma clearance of tracer to bone. The Patlak plot method was used to evaluate whole skeleton 99mTc-MDP skeletal plasma clearance (Kbone) and to derive regional values for the skull, mandible, spine, pelvis, and upper and lower extremities.
  milliliter/minute
    whole skeleton | 38.30 [33.00 to 40.90]
    skull | 3.07 [2.43 to 3.74]
    mandible | 0.17 [0.13 to 0.24]
    spine | 6.32 [4.88 to 7.00]
    pelvis | 5.92 [5.78 to 6.77]
    upper extremities | 3.70 [3.41 to 5.15]
    lower extremities | 9.12 [7.82 to 9.86]
Skeletal uptake of 99m Technetium methylene diphosphonate (99m Tc-MDP) [Median (Inter-Quartile Range); unit: percentage of uptake] — Skeletal uptake describes the percent uptake of radionuclide tracer by the skeleton. Skeletal uptake is defined as percentage of uptake of 99mTc-MDP 4 hours after injection. This value differs from skeletal plasma clearance measurements because it only quantifies the amount of 99mTc-MDP taken up by bone without consideration of concentration of tracer in the plasma.
  percentage of uptake
    whole skeleton | 29.4 [27.40 to 31.70]
    skull | 2.59 [1.96 to 2.95]
    mandible | 0.14 [0.12 to 0.19]
    spine | 4.85 [3.87 to 5.68]
    pelvis | 4.57 [4.06 to 5.28]
    upper extremities | 2.98 [2.29 to 3.81]
    lower extremities | 7.09 [6.27 to 8.46]
Weight [Mean (Standard Deviation); unit: kilogram] | 63.80 (13.56)
Years post menopause [Mean (Standard Deviation); unit: years] | 21.84 (7.65)

OUTCOME MEASURES:

1. Secondary Outcome: Change in Skeletal Plasma Clearance of 99m Technetium Methylene Diphosphonate (99m Tc-MDP) in the Whole Skeleton, Skull, Mandible, Spine, Pelvis, Upper Extremities, and Lower Extremities
Description: Skeletal plasma clearance is defined as the volume of plasma cleared of tracer (99m Tc-MDP) by the skeleton per unit time (milliliter/minute). Kbone is the rate constant representing plasma clearance of tracer to bone. The Patlak plot method was used to evaluate whole skeleton 99mTc-MDP skeletal plasma clearance (Kbone) and to derive regional values for the skull, mandible, spine, pelvis, and upper and lower extremities.
Time Frame: Baseline, 3 months, 18 months, 24 months
Population: All participants with a baseline observation and at least 1 post-baseline observation.
Measure: Median (Inter-Quartile Range); unit: percentage of change of plasma clearance
Arm/Group | Teriparatide
Number analyzed (Participants) | 10
percentage of change of plasma clearance
  Whole skeleton, baseline to 3 months, n=10 | 25.02 [14.21 to 30.73]
  Whole skeleton, baseline to 24 months, n=9 | 3.52 [-8.27 to 11.93]
  Whole skeleton, 3 months to 18 months, n=10 | 10.44 [7.83 to 21.00]
  Whole skeleton, 18 months to 24 months, n=9 | -22.20 [-24.35 to -18.39]
  Skull, baseline to 3 months, n=8 | 72.25 [42.19 to 106.56]
  Skull, baseline to 18 months, n=8 | 128.44 [97.38 to 162.55]
  Skull, baseline to 24 months, n=7 | 21.20 [8.00 to 54.90]
  Skull, 3 months to 18 months, n=8 | 31.01 [17.65 to 47.29]
  Skull, 18 months to 24 months, n=7 | -37.87 [-45.64 to -32.14]
  Mandible, baseline to 3 months, n=8 | 65.94 [26.56 to 106.76]
  Mandible, baseline to 18 months, n=8 | 60.99 [31.25 to 127.78]
  Mandible, baseline to 24 months, n=7 | 21.05 [-6.90 to 82.35]
  Mandible, 3 months to 18 months, n=8 | 4.55 [-3.25 to 15.13]
  Mandible, 18 months to 24 months, n=7 | -17.39 [-25.81 to -10.00]
  Spine, baseline to 3 months, n=10 | 17.31 [0.46 to 35.53]
  Spine, baseline to 18 months, n=10 | 33.81 [7.53 to 57.99]
  Spine, baseline to 24 months, n=9 | 16.94 [-0.14 to 32.99]
  Spine, 3 months to 18 months, n=10 | 14.10 [-0.23 to 20.00]
  Spine, 18 months to 24 months, n=9 | -9.42 [-15.31 to 8.31]
  Pelvis, baseline to 3 months, n=10 | 20.26 [5.00 to 43.59]
  Pelvis, baseline to 18 months, n=10 | 8.36 [4.15 to 28.23]
  Pelvis, baseline to 24 months, n=9 | -5.58 [-14.19 to 10.65]
  Pelvis, 3 months to 18 months, n=10 | -3.29 [-15.75 to 2.15]
  Pelvis, 18 months to 24 months, n=9 | -13.81 [-17.61 to 2.26]
  Upper extremities, baseline to 3 months, n=10 | 42.52 [8.92 to 91.09]
  Upper extremities, baseline to 18 months, n=10 | 95.49 [62.52 to 146.10]
  Upper extremities, baseline to 24 months, n=9 | 62.76 [31.07 to 70.24]
  Upper extremities, 3 months to 18 months, n=10 | 45.84 [24.27 to 77.33]
  Upper extremities, 18 months to 24 months, n=9 | -19.35 [-27.59 to 1.18]
  Lower extremities, baseline to 3 months, n=10 | 20.98 [3.71 to 50.16]
  Lower extremities, baseline to 18 months, n=10 | 34.88 [16.65 to 67.09]
  Lower extremities, baseline to 24 months, n=9 | 7.07 [-8.08 to 15.77]
  Lower extremities, 3 months to 18 months, n=10 | 12.72 [-12.14 to 24.74]
  Lower extremities, 18 months to 24 months, n=9 | -20.72 [-21.81 to -13.55]
Statistical Analysis 1: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the skull from baseline to 3 months; Test type: Superiority or Other; p = 0.0078, Wilcoxon signed rank test — p-value is for skull, baseline to 3 months
Statistical Analysis 2: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the skull from baseline to 18 months; Test type: Superiority or Other; p = 0.0078, Wilcoxon signed rank test — p-value is for skull, baseline to 18 months
Statistical Analysis 3: Comparison: Teriparatide; Tested was the hypothesis that there would be no change in skeletal plasma clearance of 99m Tc-MDP in the skull from baseline to 24 months; Test type: Superiority or Other; p = 0.0313, Wilcoxon signed rank test — p-value is for skull, baseline to 24 months
Statistical Analysis 4: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the skull from 3 months to 18 months; Test type: Superiority or Other; p = 0.0078, Wilcoxon signed rank test — p-value is for skull, 3 months to 18 months
Statistical Analysis 5: Comparison: Teriparatide; Tested was the hypothesis that there would be no decrease in skeletal plasma clearance of 99m Tc-MDP in the skull from 18 months to 24 months; Test type: Superiority or Other; p = 0.0156, Wilcoxon signed rank test — p-value is for skull, 18 months to 24 months
Statistical Analysis 6: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the mandible from baseline to 3 months; Test type: Superiority or Other; p = 0.0156, Wilcoxon signed rank test — p-value is for mandible, baseline to 3 months
Statistical Analysis 7: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the mandible from baseline to 18 months; Test type: Superiority or Other; p = 0.0078, Wilcoxon signed rank test — p-value is for mandible, baseline to 18 months
Statistical Analysis 8: Comparison: Teriparatide; Tested was the hypothesis that there would be no change in skeletal plasma clearance of 99m Tc-MDP in the mandible from baseline to 24 months; Test type: Superiority or Other; p = 0.1563, Wilcoxon signed rank test — p-value is for mandible, baseline to 24 months
Statistical Analysis 9: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the mandible from 3 months to 18 months; Test type: Superiority or Other; p = 0.4375, Wilcoxon signed rank test — p-value is for mandible, 3 months to 18 months
Statistical Analysis 10: Comparison: Teriparatide; Tested was the hypothesis that there would be no decrease in skeletal plasma clearance of 99m Tc-MDP in the mandible from 18 months to 24 months; Test type: Superiority or Other; p = 0.0781, Wilcoxon signed rank test — p-value is for mandible, 18 months to 24 months
Statistical Analysis 11: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the spine from baseline to 3 months; Test type: Superiority or Other; p = 0.0371, Wilcoxon signed rank test — p-value is for spine, baseline to 3 months
Statistical Analysis 12: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the spine from baseline to 18 months; Test type: Superiority or Other; p = 0.0137, Wilcoxon signed rank test — p-value is for spine, baseline to 18 months
Statistical Analysis 13: Comparison: Teriparatide; Tested was the hypothesis that there would be no change in skeletal plasma clearance of 99m Tc-MDP in the spine from baseline to 24 months; Test type: Superiority or Other; p = 0.0547, Wilcoxon signed rank test — p-value is for spine, baseline to 24 months
Statistical Analysis 14: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the spine from 3 months to 18 months; Test type: Superiority or Other; p = 0.0488, Wilcoxon signed rank test — p-value is for spine, 3 months to 18 months
Statistical Analysis 15: Comparison: Teriparatide; Tested was the hypothesis that there would be no decrease in skeletal plasma clearance of 99m Tc-MDP in the spine from 18 months to 24 months; Test type: Superiority or Other; p = 0.3594, Wilcoxon signed rank test — p-value is for spine, 18 months to 24 months
Statistical Analysis 16: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the pelvis from baseline to 3 months; Test type: Superiority or Other; p = 0.0488, Wilcoxon signed rank test — p-value is for pelvis, baseline to 3 months
Statistical Analysis 17: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the pelvis from baseline to 18 months; Test type: Superiority or Other; p = 0.1055, Wilcoxon signed rank test — p-value is for pelvis, baseline to 18 months
Statistical Analysis 18: Comparison: Teriparatide; Tested was the hypothesis that there would be no change in skeletal plasma clearance of 99m Tc-MDP in the pelvis from baseline to 24 months; Test type: Superiority or Other; p = 0.9102, Wilcoxon signed rank test — p-value is for pelvis, baseline to 24 months
Statistical Analysis 19: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the pelvis from 3 months to 18 months; Test type: Superiority or Other; p = 0.1934, Wilcoxon signed rank test — p-value is for pelvis, 3 months to 18 months
Statistical Analysis 20: Comparison: Teriparatide; Tested was the hypothesis that there would be no decrease in skeletal plasma clearance of 99m Tc-MDP in the pelvis from 18 months to 24 months; Test type: Superiority or Other; p = 0.1641, Wilcoxon signed rank test — p-value is for pelvis, 18 months to 24 months
Statistical Analysis 21: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the upper extremities from baseline to 3 months; Test type: Superiority or Other; p = 0.0137, Wilcoxon signed rank test — p-value is for upper extremities, baseline to 3 months
Statistical Analysis 22: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the upper extremities from baseline to 18 months; Test type: Superiority or Other; p = 0.0020, Wilcoxon signed rank test — p-value is for upper extremities, baseline to 18 months
Statistical Analysis 23: Comparison: Teriparatide; Tested was the hypothesis that there would be no change in skeletal plasma clearance of 99m Tc-MDP in the upper extremities from baseline to 24 months; Test type: Superiority or Other; p = 0.0039, Wilcoxon signed rank test — p-value is for upper extremities, baseline to 24 months
Statistical Analysis 24: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the upper extremities from 3 months to 18 months; Test type: Superiority or Other; p = 0.0273, Wilcoxon signed rank test — p-value is for upper extremities, 3 months to 18 months
Statistical Analysis 25: Comparison: Teriparatide; Tested was the hypothesis that there would be no decrease in skeletal plasma clearance of 99m Tc-MDP in the upper extremities from 18 months to 24 months; Test type: Superiority or Other; p = 0.0547, Wilcoxon signed rank test — p-value is for upper extremities, 18 months to 24 months
Statistical Analysis 26: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the lower extremities from baseline to 3 months; Test type: Superiority or Other; p = 0.0195, Wilcoxon signed rank test — p-value is for lower extremities, baseline to 3 months
Statistical Analysis 27: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the lower extremities from baseline to 18 months; Test type: Superiority or Other; p = 0.0059, Wilcoxon signed rank test — p-value is for lower extremities, baseline to 18 months
Statistical Analysis 28: Comparison: Teriparatide; Tested was the hypothesis that there would be no change in skeletal plasma clearance of 99m Tc-MDP in the lower extremities from baseline to 24 months; Test type: Superiority or Other; p = 0.5703, Wilcoxon signed rank test — p-value is for lower extremities, baseline to 24 months
Statistical Analysis 29: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the lower extremities from 3 months to 18 months; Test type: Superiority or Other; p = 0.1934, Wilcoxon signed rank test — p-value is for lower extremities, 3 months to 18 months
Statistical Analysis 30: Comparison: Teriparatide; Tested was the hypothesis that there would be no decrease in skeletal plasma clearance of 99m Tc-MDP in the lower extremities from 18 months to 24 months; Test type: Superiority or Other; p = 0.0039, Wilcoxon signed rank test — p-value is for lower extremities, 18 months to 24 months
Statistical Analysis 31: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the whole body from baseline to 3 months; Test type: Superiority or Other; p = 0.0039, Wilcoxon signed rank test — p-value is for whole body, baseline to 3 months
Statistical Analysis 32: Comparison: Teriparatide; Tested was the hypothesis that there would be no change in skeletal plasma clearance of 99m Tc-MDP in the whole body from baseline to 24 months; Test type: Superiority or Other; p = 0.5703, Wilcoxon signed rank test — p-value is for whole body, baseline to 24 months
Statistical Analysis 33: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal plasma clearance of 99m Tc-MDP in the whole body from 3 months to 18 months; Test type: Superiority or Other; p = 0.0273, Wilcoxon signed rank test — p-value is for whole body, 3 months to 18 months
Statistical Analysis 34: Comparison: Teriparatide; Tested was the hypothesis that there would be no decrease in skeletal plasma clearance of 99m Tc-MDP in the whole body from 18 months to 24 months; Test type: Superiority or Other; p = 0.0039, Wilcoxon signed rank test — p-value if for whole body, 18 months to 24 months

2. Secondary Outcome: Change in Skeletal Uptake of 99m Technetium Methylene Diphosphonate (99m Tc-MDP) in the Whole Skeleton, Skull, Mandible, Spine, Pelvis, Upper Extremities, and Lower Extremities
Description: Skeletal uptake describes the percent uptake of radionuclide tracer by the skeleton when compared to baseline or other post-baseline measures. Skeletal uptake is defined as percentage of uptake of 99mTc-MDP 4 hours after injection. This value differs from skeletal plasma clearance measurements because it only quantifies the amount of 99mTc-MDP taken up by bone without consideration of concentration of tracer in the plasma.
Time Frame: Baseline, 3 months, 18 months, 24 months
Population: All participants with a baseline observation and at least 1 post-baseline observation.
Measure: Median (Inter-Quartile Range); unit: percentage of change of skeletal uptake
Arm/Group | Teriparatide
Number analyzed (Participants) | 10
percentage of change of skeletal uptake
  whole skeleton, baseline to 3 months, n=10 | 15.63 [4.93 to 28.89]
  whole skeleton, baseline to 18 months, n=10 | 26.12 [11.81 to 37.31]
  whole skeleton, baseline to 24 months, n=9 | 5.68 [-9.86 to 8.03]
  whole skeleton, 3 months to 18 months, n=10 | 3.99 [-5.56 to 14.44]
  whole skeleton, 18 months to 24 months, n=9 | -14.54 [-19.35 to -13.41]
  skull, baseline to 3 months, n=8 | 68.27 [32.45 to 90.26]
  skull, baseline to 18 months, n=8 | 120.85 [83.57 to 137.47]
  skull, baseline to 24 months, n=7 | 26.87 [3.31 to 50.99]
  skull, 3 months to 18 months, n=8 | 23.63 [15.75 to 50.43]
  skull, 18 months to 24 months, n=7 | -34.36 [-39.86 to -28.93]
  mandible, baseline to 3 months, n=8 | 52.20 [11.01 to 77.31]
  mandible, baseline to 18 months, n=8 | 62.91 [6.25 to 118.33]
  mandible, baseline to 24 months, n=7 | 23.08 [-8.00 to 71.43]
  mandible, 3 months to 18 months, n=8 | 3.85 [-6.45 to 14.64]
  mandible, 18 to 24 months, n=7 | -6.25 [-23.81 to -4.17]
  spine, baseline to 3 months, n=10 | 12.15 [-4.45 to 21.92]
  spine, baseline to 18 months, n=10 | 17.77 [-3.76 to 40.50]
  spine, baseline to 24 months, n=9 | 17.68 [6.92 to 38.50]
  spine, 3 months to 18 months, n=10 | 13.36 [-9.34 to 29.41]
  spine, 18 months to 24 months, n=9 | -0.19 [-5.04 to 7.63]
  pelvis, baseline to 3 months, n=10 | 14.26 [-0.60 to 40.06]
  pelvis, baseline to 18 months, n=10 | -1.21 [-8.33 to 31.41]
  pelvis, baseline to 24 months, n=9 | -1.48 [-10.80 to 6.19]
  pelvis, 3 months to 18 months, n=10 | -3.70 [-18.24 to 3.47]
  pelvis, 18 months to 24 months, n=9 | -5.23 [-8.47 to 3.10]
  upper extremities, baseline to 3 months, n=10 | 31.59 [17.21 to 53.87]
  upper extremities, baseline to 18 months, n=10 | 76.58 [48.76 to 120.47]
  upper extremities, baseline to 24 months, n=9 | 57.82 [35.95 to 74.24]
  upper extremities, 3 months to 18 months, n=10 | 48.58 [25.17 to 59.96]
  upper extremities, 18 months to 24 months, n=9 | -10.13 [-18.07 to 0.40]
  lower extremities, baseline to 3 months, n=10 | 9.25 [3.64 to 54.37]
  lower extremities, baseline to 18 months, n=10 | 23.98 [10.53 to 52.89]
  lower extremities, baseline to 24 months, n=9 | 0.86 [-4.37 to 13.33]
  lower extremities, 3 months to 18 months, n=10 | 7.58 [-3.71 to 22.31]
  lower extremities, 18 months to 24 months, n=9 | -16.99 [-19.94 to -2.17]
Statistical Analysis 1: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the whole skeleton from baseline to 3 months; Test type: Superiority or Other; p = 0.0098, Wilcoxon signed rank test — p-value is for whole skeleton, baseline to 3 months
Statistical Analysis 2: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the whole skeleton from baseline to 18 months; Test type: Superiority or Other; p = 0.0039, Wilcoxon signed rank test — p-value is for whole skeleton, baseline to 18 months
Statistical Analysis 3: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the whole skeleton from baseline to 24 months; Test type: Superiority or Other; p = 0.6523, Wilcoxon signed rank test — p-value is for whole skeleton, baseline to 24 months
Statistical Analysis 4: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the whole skeleton from 3 months to 18 months; Test type: Superiority or Other; p = 0.1641, Wilcoxon signed rank test — p-value is for whole skeleton, 3 months to 18 months
Statistical Analysis 5: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the whole skeleton from 18 months to 24 months; Test type: Superiority or Other; p = 0.0078, Wilcoxon signed rank test — p-value is for whole skeleton, 18 months to 24 months
Statistical Analysis 6: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the skull from baseline to 3 months; Test type: Superiority or Other; p = 0.0078, Wilcoxon signed rank test — p-value is for skull, baseline to 3 months
Statistical Analysis 7: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the skull from baseline to 18 months; Test type: Superiority or Other; p = 0.0078, Wilcoxon signed rank test — p-value is for skull, baseline to 18 months
Statistical Analysis 8: Comparison: Teriparatide; Tested was the hypothesis that there would be no change in skeletal uptake of 99m Tc-MDP in the skull from baseline to 24 months; Test type: Superiority or Other; p = 0.0781, Wilcoxon signed rank test — p-value is for skull, baseline to 24 months
Statistical Analysis 9: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the skull from 3 months to 18 months; Test type: Superiority or Other; p = 0.0078, Wilcoxon signed rank test — p-value is for skull, 3 months to 18 months
Statistical Analysis 10: Comparison: Teriparatide; Tested was the hypothesis that there would be no decrease in skeletal uptake of 99m Tc-MDP in the skull from 18 months to 24 months; Test type: Superiority or Other; p = 0.0156, Wilcoxon signed rank test — p-value is for skull, 18 months to 24 months
Statistical Analysis 11: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the mandible from baseline to 3 months; Test type: Superiority or Other; p = 0.0391, Wilcoxon signed rank test — p-value is for mandible, baseline to 3 months
Statistical Analysis 12: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the mandible from baseline to 18 months; Test type: Superiority or Other; p = 0.0313, Wilcoxon signed rank test — p-value is for mandible, baseline to 18 months
Statistical Analysis 13: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the mandible from baseline to 24 months; Test type: Superiority or Other; p = 0.2969, Wilcoxon signed rank test — p-value is for mandible, baseline to 24 months
Statistical Analysis 14: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the mandible from 3 months to 18 months; Test type: Superiority or Other; p = 0.5625, Wilcoxon signed rank test — p-value is for mandible, 3 months to 18 months
Statistical Analysis 15: Comparison: Teriparatide; Tested was the hypothesis that there would be no decrease in skeletal uptake of 99m Tc-MDP in the mandible from 18 months to 24 months; Test type: Superiority or Other; p = 0.0469, Wilcoxon signed rank test — p-value is for mandible, 18 months to 24 months
Statistical Analysis 16: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the spine from 3 months to 18 months; Test type: Superiority or Other; p = 0.1934, Wilcoxon signed rank test — p-value is for spine, 3 months to 18 months
Statistical Analysis 17: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the spine from baseline to 3 months; Test type: Superiority or Other; p = 0.2324, Wilcoxon signed rank test — p-value is for spine, baseline to 3 months
Statistical Analysis 18: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the spine from baseline to 18 months; Test type: Superiority or Other; p = 0.0645, Wilcoxon signed rank test — p-value is for spine, baseline to 18 months
Statistical Analysis 19: Comparison: Teriparatide; Tested was the hypothesis that there would be no change in skeletal uptake of 99m Tc-MDP in the spine from baseline to 24 months; Test type: Superiority or Other; p = 0.0273, Wilcoxon signed rank test — p-value is for spine, baseline to 24 months
Statistical Analysis 20: Comparison: Teriparatide; Tested was the hypothesis that there would be no decrease in skeletal uptake of 99m Tc-MDP in the spine from 18 months to 24 months; Test type: Superiority or Other; p = 0.7344, Wilcoxon signed rank test — p-value is for spine, 18 months to 24 months
Statistical Analysis 21: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the pelvis from baseline to 3 months; Test type: Superiority or Other; p = 0.1934, Wilcoxon signed rank test — p-value is for pelvis, baseline to 3 months
Statistical Analysis 22: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the pelvis from baseline to 18 months; Test type: Superiority or Other; p = 0.7695, Wilcoxon signed rank test — p-value is for pelvis, baseline to 18 months
Statistical Analysis 23: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the pelvis from baseline to 24 months; Test type: Superiority or Other; p = 0.6523, Wilcoxon signed rank test — p-value is for pelvis, baseline to 24 months
Statistical Analysis 24: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the pelvis from 3 months to 18 months; Test type: Superiority or Other; p = 0.2324, Wilcoxon signed rank test — p-value is for pelvis, 3 months to 18 months
Statistical Analysis 25: Comparison: Teriparatide; Tested was the hypothesis that there would be no decrease in skeletal uptake of 99m Tc-MDP in the pelvis from 18 months to 24 months; Test type: Superiority or Other; p = 0.6523, Wilcoxon signed rank test — p-value is for pelvis, 18 months to 24 months
Statistical Analysis 26: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the upper extremities from baseline to 3 months; Test type: Superiority or Other; p = 0.0098, Wilcoxon signed rank test — p-value is for upper extremities, baseline to 3 months
Statistical Analysis 27: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the upper extremities from baseline to 18 months; Test type: Superiority or Other; p = 0.0020, Wilcoxon signed rank test — p-value is for upper extremities, baseline to 18 months
Statistical Analysis 28: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the upper extremities from baseline to 24 months; Test type: Superiority or Other; p = 0.0039, Wilcoxon signed rank test — p-value is for upper extremities, baseline to 24 months
Statistical Analysis 29: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the upper extremities from 3 months to 18 months; Test type: Superiority or Other; p = 0.0273, Wilcoxon signed rank test — p-value is for upper extremities, 3 months to 18 months
Statistical Analysis 30: Comparison: Teriparatide; Tested was the hypothesis that there would be no decrease in skeletal uptake of 99m Tc-MDP in the upper extremities from 18 months to 24 months; Test type: Superiority or Other; p = 0.3594, Wilcoxon signed rank test — p-value is for upper extremities, 18 months to 24 months
Statistical Analysis 31: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the lower extremities from baseline to 3 months; Test type: Superiority or Other; p = 0.0371, Wilcoxon signed rank test — p-value is for lower extremities, baseline to 3 months
Statistical Analysis 32: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the lower extremities from baseline to 18 months; Test type: Superiority or Other; p = 0.0098, Wilcoxon signed rank test — p-value is for lower extremities, baseline to 18 months
Statistical Analysis 33: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the lower extremities from baseline to 24 months; Test type: Superiority or Other; p = 0.4609, Wilcoxon signed rank test — p-value is for lower extremities, baseline to 24 months
Statistical Analysis 34: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in skeletal uptake of 99m Tc-MDP in the lower extremities from 3 months to 18 months; Test type: Superiority or Other; p = 0.1934, Wilcoxon signed rank test — p-value is for lower extremities, 3 months to 18 months
Statistical Analysis 35: Comparison: Teriparatide; Tested was the hypothesis that there would be no decrease in skeletal uptake of 99m Tc-MDP in the lower extremities from 18 months to 24 months; Test type: Superiority or Other; p = 0.0273, Wilcoxon signed rank test — p-value is for lower extremities, 18 months to 24 months

3. Secondary Outcome: Change in Qualitative Visual Scores of Focal Uptake of 99m Technetium Methylene Diphosphonate (99m Tc-MDP) in the Whole Skeleton
Description: Changes in focal uptake (localized, defined areas of uptake) were visually scored and compared to baseline or other post-baseline assessments. Changes were rated on a scale from 0-4: 0=no clinically significant focal areas of skeletal uptake; 1=focal areas affecting <1% of skeleton; 2=focal areas affecting >=5% of skeleton; 3=focal areas affecting >=20% of skeleton; 4=focal areas affecting >=50% of skeleton.
Time Frame: Baseline, 3 months, 18 months, 24 months
Population: All participants with a baseline observation and at least 1 post-baseline observation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teriparatide
Number analyzed (Participants) | 10
units on a scale
  focal change, baseline to 3 months, n=10 | 0.1 (0.32) [0 to 0]
  focal change, baseline to 18 months, n=10 | 0.1 (0.32) [0.0 to 0.0]
  focal change, baseline to 24 months, n=9 | 0 (0) [0 to 0]
  focal change, 3 months to 18 months, n=10 | 0 (0) [0 to 0]
  focal change, 18 months to 24 months, n=9 | 0 (0) [0 to 0]
Statistical Analysis 1: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in focal skeletal uptake of 99m Tc-MDP from baseline to 3 months; Test type: Superiority or Other; p = 1.0, Wilcoxon signed rank test — p-value is for focal change, baseline to 3 months
Statistical Analysis 2: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in focal skeletal uptake of 99m Tc-MDP from baseline to 18 months; Test type: Superiority or Other; p = 1.0, Wilcoxon signed rank test — p-value is for focal change, baseline to 18 months

4. Secondary Outcome: Number of Participants With Changes in Diffuse Uptake of 99m Tc-MDP - Qualitative Visual Assessment in the Whole Skeleton
Description: Changes in diffuse uptake were determined by comparing diffuse uptake to baseline or other post-baseline observations. Diffuse uptake indicates response to therapy (during active treatment, increased diffuse uptake was expected; after the 6-month withdrawal period, decreased diffuse uptake was expected). Qualitative visual scoring of changes in the bone scan images were performed jointly by 3 reviewers who classified changes in the whole skeleton into 4 groups as follows: possible decreased response, no response, possible response, and definite response.
Time Frame: baseline, 3 months, 18 months, 24 months
Population: All participants with a baseline observation and at least 1 post-baseline observation.
Measure: Number; unit: participants
Arm/Group | Teriparatide
Number analyzed (Participants) | 10
participants
  3 months, no response | 2
  3 months, possible response | 2
  3 months, definite response | 6
  18 months, no response | 1
  18 months, possible response | 1
  18 months, definite response | 8
  24 months, possible response | 1
  24 months, no response | 6
  24 months, possible response | 1
  24 months, definite response | 1

5. Primary Outcome: Change From Baseline in Whole Skeleton Skeletal Plasma Clearance of 99m Technetium Methylene Diphosphonate (99m Tc-MDP) to 18 Months
Description: Skeletal plasma clearance is defined as the volume of plasma cleared of tracer (99m Tc-MDP) by the skeleton per unit time (milliliter/minute). Kbone is the rate constant representing plasma clearance of tracer to bone. The Patlak plot method was used to evaluate whole skeleton 99mTc-MDP skeletal plasma clearance (Kbone).
Time Frame: baseline, 18 months
Population: All participants with a baseline observation and at least 1 post-baseline observation.
Measure: Median (Inter-Quartile Range); unit: percentage of change of plasma clearance
Arm/Group | Teriparatide
Number analyzed (Participants) | 10
percentage of change of plasma clearance | 33.75 [29.97 to 50.91]
Statistical Analysis 1: Comparison: Teriparatide; Tested was the hypothesis that there would be no increase in whole skeletal plasma clearance of 99m Tc-MDP from baseline to 18 months; Test type: Superiority or Other; p = 0.0020, Wilcoxon signed rank test — p-value is for change at 18 months

ADVERSE EVENTS:
Arm/Group | Teriparatide
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=12)
Chest pain (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=12)
Arrhythmia (Cardiac disorders) | 2 (3)
Palpitations (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 1 (1)
Eustachian tube obstruction (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (2)
Blepharitis (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Chorioretinal disorder (Eye disorders) | 1 (1)
Optic atrophy (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Lip disorder (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Chest pain (General disorders) | 2 (2)
Cyst (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Feeling hot (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (2)
Injection site haematoma (General disorders) | 1 (3)
Injection site irritation (General disorders) | 1 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (3)
Kidney infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Fractured coccyx (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood pressure increased (Investigations) | 2 (2)
Cardiac murmur (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (2)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (4)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Extensor plantar response (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Lethargy (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Nerve compression (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days